CLINICAL TRIAL: NCT00002205
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Amprenavir (141W94) and Abacavir Combination Therapy in Protease Inhibitor Experienced Subjects With HIV-1 Infection Who Are Failing Their Current Antiretroviral Treatment Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 264H
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: HIV Protease Inhibitors; VX 478; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — abacavir; amprenavir

INTERVENTIONS:
Drug: Abacavir sulfate
Drug: Amprenavir

SUMMARY:
To assess the safety, tolerance, and efficacy of amprenavir (APV) plus abacavir (ABC) in patients who have previously failed antiretroviral treatment containing a protease inhibitor (PI). To provide open-label, pre-approval access to APV for adults and adolescents with HIV-1 infection and limited treatment options.

This study is being conducted to provide open-label APV to patients in danger of HIV disease progression, as well as those who may benefit beyond the expected outcomes of current anti-retroviral therapies. Despite unapproved status, APV may prove highly efficacious in combatting HIV progression and may help those in need, prior to regulatory approval.

DETAILED DESCRIPTION:
This study is being conducted to provide open-label APV to patients in danger of HIV disease progression, as well as those who may benefit beyond the expected outcomes of current anti-retroviral therapies. Despite unapproved status, APV may prove highly efficacious in combatting HIV progression and may help those in need, prior to regulatory approval.

Patients are stratified into one of the following treatment options:

Non-nucleoside reverse transcriptase inhibitor (NNRTI)-naive:

Option 1- APV / ABC / PI / NNRTI / +nucleoside reverse transcriptase inhibitor(s) (NRTI) Option 2- APV / ABC / NNRTI / NRTI(s)

NNRTI-Experienced Patients:

Option 1- APV / ABC / PI / +NRTI(s) Option 2- APV / ABC / +NRTI(s) To assess clinical efficacy, lab values (i.e., hematology, serum chemistry, plasma HIV-1 viral load determination and CD4+ cell count measurements) are collected at pre-entry and every 12 weeks thereafter.

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Hepatic failure with elevated ALT and AST values.
* Malabsorption syndrome or other gastrointestinal dysfunction which may interfere with drug absorption or render the patient unable to take oral medication.
* Renal failure requiring dialysis.

Concurrent Medication:

Excluded:

Patients currently participating in, or who would qualify for or have access to, an enrolling study of APV (ACTG 398 and ACTG 400).

Patients with the following prior conditions are excluded:

* Patients suffering from serious medical conditions such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction which, in the opinion of the investigator, would compromise the safety of the patient.
* History of clinically relevant pancreatitis or hepatitis within the last 6 months.

Prior Medication:

Excluded:

* Previous treatment with more than one HIV protease inhibitor.
* ABC use for greater than 8 weeks prior to enrollment into this study.

Risk Behavior:

Excluded:

Patients with current alcohol or illicit drug use which, in the opinion of the investigator, would interfere with the patient's ability to comply with the requirements of the study.

Patients have:

* HIV-1 infection.
* CD4+ cell count less than or equal to 400 cells/mm3 and plasma HIV-1 RNA greater than or equal to 10,000 copies/ml at the first pre-entry assessment.
* Evidence of failure on an antiretroviral treatment regimen containing a protease inhibitor.
* Clinical evidence of failure in their current regimen and require antiretroviral therapy, and need APV plus ABC to induce viral load suppression.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Glaxo Wellcome Inc, Research Triangle Park, North Carolina, United States